CLINICAL TRIAL: NCT03303144
Title: Equivalence of Triferic® (Ferric Pyrophosphate Citrate) Administered Via Hemodialysate and Intravenously to Adult CKD-5HD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-20
Record Dates: First submitted 2017-09-28; First posted 2017-10-05 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: End Stage Renal Disease
Keywords: Pharmacokinetics; Equivalence
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Triferic via Hemodialysate (Experimental): Triferic will be mixed with the liquid bicarbonate concentrate used in the preparation of the hemodialysate solution. This will result in a final Triferic iron concentration in the dialysate of 2 µM (110 µg/L). The patients will receive Triferic over 4 hrs at one hemodialysis session.
  Interventions: Drug: Triferic
- Triferic via IV infusion( pre-dialyzer) (Experimental): Patients will receive a single 6.5-mg dose of Triferic iron administered IV over 3 hrs during hemodialysis via arterial blood line (pre-dialyzer)
  Interventions: Drug: Triferic
- Triferic via IV infusion (post-dialyzer) (Experimental): Patients will receive a single 6.5-mg dose of Triferic iron administered IV over 3 hrs during hemodialysis via venous blood line (post-dialyzer)
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic — ferric pyrophosphate citrate
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
The main purpose is to establish the equivalence of Triferic iron administered via dialysate into the arterial blood line and into the venous blood line

DETAILED DESCRIPTION:
An open-label, four period, randomized, crossover study of Triferic iron administered via hemodialysis compared to Triferic administered intravenously pre- and post- hemodialyzer.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to provide informed consent and have personally signed and dated the written informed consent document before completing any study-related procedures.
2. The patient must be 18-80 years of age inclusive at the time of consent.
3. The patient must have been undergoing chronic hemodialysis for chronic kidney disease for at least 3 months, and be expected to remain on hemodialysis and be able to complete the study.
4. The patient must have a Screening ferritin level of ≥100µg/L.
5. The patient must have a Screening transferrin saturation (TSAT) of 15-45%, inclusive.
6. The patient must have a Screening hemoglobin (Hgb) concentration ≥9.0 g/dL.
7. The patient must be undergoing hemodialysis at least 3x/week.
8. The patient must have at least a minimally adequate measured dialysis dose defined as single-pool Kt/V (dialyzer clearance of urea multiplied by dialysis time, divided by patient's total body water) ≥1.2, or KIDt/V (online dialyzer clearance measured using ionic dialysance multiplied by dialysis time, divided by patient's total body water) ≥1.2 measured within the 90 days prior to HD #1.
9. Patient is receiving, or can receive anticoagulation for dialysis by a single dose of unfractionated heparin or low molecular weight heparin pre-dialysis; or by intermittent IV heparin bolus.
10. The patient's vascular access for dialysis that will be used during the study must have stable function in the judgment of the Investigator.
11. The patient must agree to discontinue all iron preparations (oral and IV) for 14 days prior to the start of HD#1 and throughout the study.
12. Female patients must not be pregnant or breastfeeding. They must have been amenorrheic for the past year or be surgically sterile or agree to not become pregnant by continuous use of an effective birth control method acceptable to the Investigator for the duration of their participation in the study.

Exclusion Criteria:

1. The patient has had an RBC or whole blood transfusion within 4 weeks prior to Screening.
2. The patient requires a continuous infusion of heparin during standard hemodialysis.
3. The patient has had administration of IV or oral iron supplements (including multivitamins with iron or iron based phosphate binders) within 14 days prior to the start of HD #1. (The patient may subsequently become eligible if additional time elapses and all other eligibility criteria are met.).
4. The patient has known active bleeding from any site other than AV fistula or graft (e.g., gastrointestinal, hemorrhoidal, nasal, pulmonary, etc.).
5. The patient has a living kidney donor identified or living-donor kidney transplant scheduled to occur during study participation. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
6. The patient is scheduled to have a surgical procedure during the study.
7. The patient has had a hospitalization within the 4 weeks prior to Screening (except for vascular access surgery) that, in the opinion of the Investigator, confers a significant risk of hospitalization during the course of the study.
8. The patient has a history of noncompliance with the dialysis regimen in the opinion of the Investigator.
9. The patient has a known ongoing active inflammatory disorder (other than CKD), such as systemic lupus erythematosus, rheumatoid arthritis, or other collagen-vascular disease, that currently requires systemic anti-inflammatory or immunomodulatory therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 27 participants in the study were randomly assigned to cross-over between the three treatments on Day 3, Day 8 and Day 10.
Groups:
- Triferic Via Hemodialysate (Day 3): Triferic will be mixed with the liquid bicarbonate concentrate used in the preparation of the hemodialysate solution. This will result in a final Triferic iron concentration in the dialysate of 2 µM (110 µg/L). The patients will receive Triferic over 4 hrs at one hemodialysis session.
- Triferic Via IV Infusion( Pre-dialyzer) (Day 8): Patients will receive a single 6.5-mg dose of Triferic iron administered IV over 3 hrs during hemodialysis via arterial blood line (pre-dialyzer)
- Triferic Via IV Infusion (Post-dialyzer) (Day 10): Patients will receive a single 6.5-mg dose of Triferic iron administered IV over 3 hrs during hemodialysis via venous blood line (post-dialyzer)
Period: Triferic Via Hemodialysate (Day 3)
Arm/Group | Triferic Via Hemodialysate (Day 3) | Triferic Via IV Infusion( Pre-dialyzer) (Day 8) | Triferic Via IV Infusion (Post-dialyzer) (Day 10)
Started | 26 | 0 | 0
Completed | 26 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Triferic Via IV Infusion (Day 8)
Arm/Group | Triferic Via Hemodialysate (Day 3) | Triferic Via IV Infusion( Pre-dialyzer) (Day 8) | Triferic Via IV Infusion (Post-dialyzer) (Day 10)
Started | 0 | 26 | 0
Completed | 0 | 25 | 0
Not Completed | 0 | 1 | 0
Period: Triferic Via IV Infusion (Day 10)
Arm/Group | Triferic Via Hemodialysate (Day 3) | Triferic Via IV Infusion( Pre-dialyzer) (Day 8) | Triferic Via IV Infusion (Post-dialyzer) (Day 10)
Started | 0 | 0 | 26
Completed | 0 | 0 | 25
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All patients in study
Arm/Group | Safety Population
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered Via Hemodialysate in Adult CKD-5HD Patients: Cmax.
Description: The PK will be done by assessing the mean Cmax of total serum iron from Triferic administered via hemodialysate, compared to Triferic administered at a fixed IV dose of 6.6 mg iron/kg during a single dialysis session.
Time Frame: 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/dL
Arm/Group | Triferic Via Hemodialysate
Number analyzed (Participants) | 25
h*ug/dL | 207 (30.4)

2. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Adult CKD-5HD Patients:Cmax
Time Frame: 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/dL
Arm/Group | Triferic Via IV Infusion( Pre-dialyzer) | Triferic Via IV Infusion (Post-dialyzer) | Triferic Via Hemodialysate
Number analyzed (Participants) | 26 | 25 | 25
h*ug/dL | 215 (21.6) | 195 (25.6) | 207 (30.4)

3. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Adult CKD-5HD Patients: AUC(0-end).
Description: The PK will be done by assessing the mean AUC(0-end) of total serum iron from Triferic administered via hemodialysate, compared to Triferic administered at a fixed IV dose of 6.5 mg iron/kg during a single dialysis session.
Time Frame: 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/dL
Arm/Group | Triferic Via IV Infusion( Pre-dialyzer) | Triferic Via IV Infusion (Post-dialyzer) | Triferic Via Hemodialysate
Number analyzed (Participants) | 26 | 25 | 25
h*ug/dL | 1540 (28.5) | 1450 (31.4) | 1500 (31.7)

4. Secondary Outcome: Safety Endpoint: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs) Incidence of Treatment Emergent Serious Adverse Events
Description: Safety will be documented by recording the incidence of treatment-emergent serious adverse events (TESAEs).The number of patients that experienced treatment emergent serious adverse events will be quantified. Please see the adverse event table for specifics.
Time Frame: From the start of the HD #1 through the end of study participation or 7 days after the last dose of Triferic, whichever is later, assessed up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Triferic Via IV Infusion( Pre-dialyzer) | Triferic Via IV Infusion (Post-dialyzer) | Triferic Via Hemodialysate
Number analyzed (Participants) | 27 | 27 | 27
Participants | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded on the AE CRF from the start of HD #1 (Day 1) through the end of study participation or 7 days after the last dose of Triferic (Day 10).
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion( Pre-dialyzer) | Triferic Via IV Infusion (Post-dialyzer)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/27 | 0/27
Other Adverse Events (participants affected / at risk) | 1/27 | 0/27 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triferic Via Hemodialysate (N=27) | Triferic Via IV Infusion( Pre-dialyzer) (N=27) | Triferic Via IV Infusion (Post-dialyzer) (N=27)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triferic Via Hemodialysate (N=27) | Triferic Via IV Infusion( Pre-dialyzer) (N=27) | Triferic Via IV Infusion (Post-dialyzer) (N=27)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03303144/Prot_SAP_000.pdf